CLINICAL TRIAL: NCT02376127
Title: Evaluation of Metastatic Spinal Bone Marrow Response to Radiation Therapy Using T1 Weighted Dynamic Contrast-Enhanced Perfusion
Brief Title: Metastatic Spinal Bone Marrow Response to Radiation Therapy Using T1 Weighted Dynamic Contrast-Enhanced Perfusion
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-203
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Solid Cancer; Metastatic Spinal Lesions
Keywords: Dynamic Contrast-Enhanced Perfusion; 14-203

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- pts with known spinal metastases: (20 patients from any solid cancer) who are to undergo radiation treatment (RT) will be recruited. The patients will undergo DCE-MRI before and after RT. RT will be classified as success based on evidence of tumor contraction on conventional MRIs, negative PET, or stability for more than 11 months and blinded from DCE MRI sequencing. For each patient, a scanning profile for the first scan will be saved and used for the follow-up scans to acquire the same locations over time. Each patient will be scanned 4 times (one pre-treatment and 3 follow up post treatment) during their consecutive clinical visits. The DCE MRI sequence is a part of MR sequences for standard care. No additional scans will be added in the standard clinical sequences.
  Interventions: Procedure: Dynamic contrast enhancement MRI

INTERVENTIONS:
Procedure: Dynamic contrast enhancement MRI

SUMMARY:
The purpose of this study is to assess imaging methods including Dynamic Contrast Enhanced Magnetic Resonance Imaging (DCE-MRI) and perfusion for the cancer that has spread to the spine. The study aims to see if using these methods will help better see response to treatment with radiation in patients with spine metastases from any solid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older
* Known pathological diagnosis of any solid cancer.
* Metastatic spinal lesions 1 cm or greater in diameter.
* Patients who are already eligible for and are to be treated with hypofractionated or single dose radiation for their spinal lesions.

Note: The patients must have their treatments at MSKCC.

Exclusion Criteria:

* Patients with renal failure or history of allergic reaction to Gadavist will be excluded.
* Patients who would be normally excluded from undergoing an MRI examination as per Memorial Hospital for Cancer and Allied Disease Screening Questionnaire for MRI.
* Patients with a pacemaker, aneurysm clip or any other condition that would warrant avoidance of a strong magnetic field.
* Patients with inability to cooperate for an MRI exam due to claustrophobia or high levels of anxiety.
* Female patients who are pregnant or nursing.
* Patients with eGFR < 30 are not eligible to higher risk of NSF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
response to treatment | 2 years
  will be based on clinical assessment and conventional MRI and PET imaging, evaluating images for evidence of tumor contraction and stable disease for more than 11 months. Clinical assessment is done by radiation oncology and is based on physical examination, patient symptoms and consideration of radiological studies.

CONTACTS AND LOCATIONS:
Overall Officials: Sasan Karimi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/